CLINICAL TRIAL: NCT06651892
Title: The Efficacy and Safety of Diluted Oral Phosphate Enema Versus Intravenous Sodium Glycerophosphate in The Treatment of Hypophosphatemia in ICU Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC #270
Record Dates: First submitted 2024-05-12; First posted 2024-10-22 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-05

CONDITIONS: Acute Hypophosphatemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - oral diluted phosphate enema (Experimental): oral diluted phosphate enema
  Interventions: Drug: Enema Phosphates Sodium
- Group B - intravenous sodium glycerophosphate (Active Comparator): intravenous sodium glycerophosphate
  Interventions: Drug: Glycophos Injectable Product

INTERVENTIONS:
Drug: Enema Phosphates Sodium — oral diluted phosphate enema containing as a repletion strategy to replace phosphate in critically ill patients with acute hypophosphatemia.
  Other Names: oral diluted phosphate enema
  Arms: Group A - oral diluted phosphate enema
Drug: Glycophos Injectable Product — intravenous sodium glycerophosphate as the standard of care or active control
  Other Names: intravenous sodium glycerophosphate
  Arms: Group B - intravenous sodium glycerophosphate

SUMMARY:
The goal of this clinical trial is to study the efficacy and safety of diluted phosphate enema in treating hypophosphatemia in adults in critical care unit in comparison to intravenous sodium glycero-phosphate as the current standard of care.

The main question it aims to answer is:

can the investigators rely on phosphate enemas as an effective and safe treatment option for hypophosphatemia in critically ill adults, in the era of global shortage of parenteral nutrition solutions and the absence of defined guidelines for treatment of acute hypophosphatemia in those population.

DETAILED DESCRIPTION:
A Randomized Controlled Trial - Non inferiority trial of 2 groups, Eligible participants will be randomly assigned to one of two groups (Intervention Group will receive Diluted Oral phosphate enema as the repletion strategy, while Control Group will receive The Standard of care: intravenous sodium glycerophosphate) for the purpose of treatment of hypophosphatemia in critically ill patients.

Dose Calculation: as per hospital protocol and scientific reference(Crook, 2009) 0.32 mmol per kg for mild hypophosphatemia 0.64 mmol per kg for moderate hypophosphatemia

All participants will be reassessed the next day after the intervention and followed up for the occurrence of any side effects, then participants will be followed up again the day after. (Assessment of serum phosphate and sodium along with occurrence of diarrhea or any other side effects).

ELIGIBILITY:
Inclusion Criteria:

* Critically ill Patients with mild (2-2.4 mg/dl) to moderate (1.5-1.9 mg/dl) hypophosphatemia.
* Serum phosphorus level less than 2.5mg/dl - between 1.5 - 2.5mg/dl
* Patients 18 years or older

Exclusion Criteria:

* Severe hypophosphatemia
* Serum Phosphorus level less than 1.5 mg/dL
* Patients on Non-peroral status
* Ileus (as paralytic ileus, post-operative)
* Any problem in gut integrity as (intestinal obstruction, Severe Malabsorption, severe diarrhea)
* Any form of ischemic gut (as mesenteric ischemia, mesenteric gastric occlusion, arterial venous insufficiency)
* Hemodynamically unstable patients
* Severe Hypocalcemia or Hypercalcemia at the beginning of the study (when iv phosphate is deemed inappropriate at the discretion of attending physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
efficacy in replacing phosphate | 2 days
  percentage of patients achieving a normal (>/=2.5mg/dl) or increase in serum level of phosphate

SECONDARY OUTCOMES:
occurrence of potential side effects | 2 days
  Monitoring of Clinical complications of phosphate replacement like diarrhea, measured as Number of events (watery diarrhea) > 3 times/day, and New Onset of Hypocalcemia /Hypercalcemia or Hypernatremia

CONTACTS AND LOCATIONS:
Locations (1):
- Al haram Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Najdi H, Sayed R, Mettawi AS, El-Hamamsy M. The efficacy and safety of diluted oral phosphate enema versus intravenous sodium glycerophosphate in the treatment of hypophosphatemia in intensive care unit patients - A non-inferiority trial. Clin Nutr ESPEN. 2025 Dec;70:692-700. doi: 10.1016/j.clnesp.2025.11.015. Epub 2025 Nov 14. PMID 41242387